CLINICAL TRIAL: NCT05687006
Title: Accuracy of Deep Inferior Epigastric Artery Perforator Mapping - Color Doppler Ultrasound Versus CT Angiography: A Randomized Controlled Trial
Brief Title: Accuracy of Deep Inferior Epigastric Artery Perforator Mapping - Color Doppler Ultrasound Versus CT Angiography
Acronym: CDUxCTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CDU2021
Record Dates: First submitted 2022-12-29; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Mammaplasty
Keywords: CT Angiography; Mammaplasty; Ultrasonography; Doppler

STUDY DESIGN:
Intervention Model Description: Randomization was carried out using an envelope method, during which the patients were randomly assigned in a ratio 1:1 to an active comparator group: "CTA+CDU (preoperative examination of vascular anatomy by CTA supplemented with vessel calibre examination of the perforator using CDU)" or an experimental group: "CDU (preoperative examination of vascular anatomy by colour duplex sonography only)".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The CTA+CDU Group (No Intervention): Every patient included in the CTA+CDU group preoperatively underwent CT angiography of the abdominal wall. Based on the CTA examination XY coordinates of DIEA perforators localized within the area between 2 cm cranial and 10 cm caudal from the umbilicus and with a vessel calibre of more than 1 mm were determined. The day before the surgery, the main perforators were marked on the patient's abdomen according to the coordinates deducted from the CTA. These perforators were additionally examined using a LOGIQ S8/V1 CDU device with a linear transducer of frequency 4-11 MHz. Any additional perforators were marked nor have CTA deducted XY coordinates of marked perforators changed based on the CDU examination. The same sonography surgeon performed all CDU examinations. The time duration of the CDU examination was measured.
- The CDU Group (Experimental): All patients included in the CDU group were examined a day before the surgery with the same CDU device by the same sonography surgeon as patients included in CTA + CDU group. During the examination, DIEA perforators were mapped and the following parameters were monitored: 1) XY coordinates of DIEA perforators localized within the area between 2 cm cranial and 10 cm caudal from the umbilicus and with a vessel calibre of more than 1 mm; 2) calibres of perforator arteries and veins; 3) PSV in the perforator artery [cm/s]; 4) velocity in the perforator vein [cm/s]; 5) the thickness of the subcutaneous tissue of the lower abdomen measured 4 cm caudal and lateral to the umbilicus. The time duration of the CDU examination was measured.
  Interventions: Procedure: Colour Doppler Ultrasound

INTERVENTIONS:
Procedure: Colour Doppler Ultrasound — The main perforators were examined using a LOGIQ S8/V1 CDU device (GE Healthcare, Chalfont St Giles, Great Britain) with a linear transducer of frequency 4-11 MHz. Measured parameters were: 1) calibre of artery and vein; 2) Peak systolic velocity (PSV) of blood in the artery [cm/s]; 3) blood velocity in the perforator vein [cm/s]; 2) the thickness of the subcutaneous tissue of the lower abdomen measured 4 cm caudal and lateral to the umbilicus. Any additional perforators were marked nor have CTA deducted XY coordinates of marked perforators changed based on the CDU examination. The same sonography surgeon performed all CDU examinations. The time duration of the CDU examination was measured.
  Other Names: CDU
  Arms: The CDU Group

SUMMARY:
The goal of this clinical trial is to compare the accuracy and contribution of Color Doppler Ultrasound (CDU) guided Deep Inferior Epigastric Artery (DIEA) perforator mapping with or without mapping using Computer Tomography angiography (CTA) in women over 18 years undergoing 2021 unilateral or bilateral breast reconstruction with an abdominal free flap.

Participants underwent scheduled reconstruction of one or both breasts with a free flap transferred from the lower abdomen. If there is a comparison group: Researchers compared interventional groups - examined using preoperative CTA of the abdominal wall supplemented with an examination of the perforators using CDU (active comparator group), and examined exclusively by using the CDU (experimental group), to see the comparison of the accuracy and contribution of CDU-guided DIEA perforator mapping with CTA mapping.

The hypothesis is that CDU examination alone is not inferior to CTA examination supplemented with parameters that CTA does not show (flow velocity, vessel diameters), by measuring these parameters with CDU.

The main questions it aims to answer are:

* To evaluate the comparison of the accuracy of surgeon-conducted CDU perforator mapping in defining the significant/dominant perforators and their exact location [XY coordinates] with the accuracy of CTA mapping.
* To compare the time duration of the CDU examination was measured.
* To measure the Fat Necrosis of the flap [3 months postoperative ]
* To measure the Flap Loss [1-week post-op, 2 weeks post-op, 6-8 weeks post-op and 3 months post-op].

DETAILED DESCRIPTION:
A blinded, randomized, prospective clinical trial was performed involving women over 18 years undergoing 2021 unilateral or bilateral breast reconstruction with an abdominal free flap. The inclusion of the mapping of major perforators as a part of preoperative deep inferior epigastric perforator (DIEP) flap planning reduces the operating time and complication rate. According to recent meta-analyses computed tomographic angiography (CTA) brings the most advantages; however, only a few studies comprising colour Doppler ultrasonography (CDU) were included with several biases in addition. Especially, studies directly comparing CTA and CDU (surgeons conducted in one study only, in one case) are rare. Recently, CDU has seen significant advances in quality and imaging capabilities, and ultrasound devices are widely available.

Women were originally randomized 1:1 to the groups one of which will undergo only CDU perforator mapping (experimental group) and the other using CTA+CDU (active comparator group). Every patient included in the CTA+CDU group preoperatively underwent CT angiography of the abdominal wall. Based on the CTA examination XY coordinates of DIEA perforators with a vessel calibre of 1 mm were determined.

The velocity and vessel diameters of these perforators were additionally examined using a CDU device. Any additional perforators were marked, nor were CTA deducted XY coordinates of marked perforators changed, based on the CDU examination. The same sonography surgeon performed all CDU examinations.

All patients included in the CDU group were examined with the same CDU device by the same sonography surgeon as patients included in CTA + CDU group. During the examination, DIEA perforators were mapped and those with a vessel calibre of 1 mm were marked and XY coordinates deducted. Calibres and velocities of perforator vessels and the abdominal subcutaneous tissue thickness were measured.

In the CTA+CDU group, CDU was used only to determine the additional parameters necessary to define categories 1-3 (according to the number of perforators). Based on CDU, coordinates were not measured in the CTA+CDU group. The main aim of this clinical study is to compare the accuracy of perforator localization (coordinates) using CDU vs. CTA.

Based on the preoperative mapping, all patients in both groups were assigned a category for each flap as follows:

A) At least one perforator of the flap meets the criteria defined for a dominant perforator. In such a case, the tactic was to dissect a single perforator flap.

B) Any perforator meets the criteria defined for a dominant perforator, but at least two perforators on the same DIEA branch meet the criteria for a significant perforator. In such a case, the tactic was to dissect the flap with the pedicle of two of those perforators.

C) Any perforator meets the criteria defined for a dominant perforator or significant perforator. In such a case, the surgical tactic was to dissect the flap with a pedicle of three perforators or as an MS-TRAM flap.

The operating surgeon was fully informed of the results of the preoperative examination and the recommended perforator or perforator selected for the flap's pedicle. However, these recommendations were not binding, and the surgeon chose the tactics of the operation taking into consideration his clinical experience. Participating in the project did not change the surgical technique and the surgery was performed as standard according to current knowledge of medicine and common practice of the department. The surgery itself was not the subject of the research. XY coordinates and diameters of the dissected perforators were measured during the surgery.

R 4.1.3 software and Joinpoint Regression 4.9.0.0. were used to perform data management and exploratory statistical analysis (p = 0.05). A two-sided Wilcoxon test was used for verification of both patient groups' comparability. The same test was used to compare the length of the CDU examination in both groups. The breaking point on the curve showing the length of the CDU examination depending on the numerical order of the examined patient was searched using the Joinpoint Regression as a secondary outcome. Euclidean distance was used to determine the difference between the CDU/CTA and during the surgery measured coordinates of the dissected perforators. Statistical testing of the difference between the accuracy of CTA and CDU examinations was performed using the GLS method. The GEE model was used to determine the difference between the CDU/CTA+CDU recommended and finally dissected a number of perforators supplying the flap.

ELIGIBILITY:
Inclusion Criteria:

* female;
* aged 18 to 65 years;
* undergoing uni- or bilateral breast free flap reconstruction harvested from the lower abdomen;
* signed informed consent to participate in the study.

Exclusion Criteria:

* history of allergy to iodinated contrast material;
* history of abdominoplasty;
* Body Mass index > 35;
* active oncological disease ;
* Karnofsky Performance Status < 50;
* change of the reconstructive method as a result of the preoperative mapping;
* non-standard performed CTA examination.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing uni- or bilateral breast-free flap reconstruction harvested from the lower abdomen.
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The average deviations (Δ) in localization of perforators in each of the groups [cm] | Through study completion, an average of 1 year
  In CDU group ΔCDU calculated for each dissected perforator as the Euclidean distance between (before the surgery, using CDU) mapped XY coordinates and the reference XY coordinates measured during the surgery. XY[0;0]=umbilicus
  In CTA+CDU group ΔCTU (because XY coordinates in this group are deducted only based on CTA, CDU in this group is used only as an additional modality to help predict the dissection category A, B, C not to deduct XY coordinates) calculated for each dissected perforator as the Euclidean distance between (before the surgery, using CTA) mapped XY coordinates and the reference XY coordinates measured during the surgery. XY[0;0]=umbilicus
The success rate in estimating proper dissecting strategy [%] | Through study completion, an average of 1 year
  In what percentage of cases the finally dissected flap category (A, B, C) is the same as the category estimated before the surgery based on CDU or CTA+CDU mapping.

SECONDARY OUTCOMES:
The time duration of the CDU examination. | 3 months post-operative
  The time duration of the CDU examination was measured.
Fat Necrosis of the flap | 3 months post-operative
  Detected using clinical examination. Assessment for fat necrosis took place 3 months postoperatively by another plastic surgeon who was therefore blinded to the mapping method.
Flap Loss | 1 week post-op, 2 weeks post-op, 6-8 weeks post-op and 3 months post-op
  Partial flap loss defined as tissue loss greater than 5 percent of the flap or clinically manifested fat necrosis. Total flap loss was also assessed. These assessments were done during regular follow-up appointments with the care team.

CONTACTS AND LOCATIONS:
Overall Officials: Libor Streit, MD, PhD., Principal Investigator — St. Anne´s University Hospital Brno
Locations (1):
- St. Anne´s University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No